CLINICAL TRIAL: NCT04678128
Title: Dance4Healing: a Pilot Study to Explore the Benefits of Tele-Dance in Individuals with an Implantable Cardioverter Defibrillator
Brief Title: Dance4Healing: Explore the Benefits of Tele-Dance in Individuals with an Implantable Cardioverter-defibrillator (ICD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to establish contract with Dance For Healing platform, so had to withdraw study
Sponsor: Sanjiv Narayan, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB # 58348
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: ICD; Anxiety; Patient Engagement
Keywords: ICD; Anxiety; QOL; Engagement
MeSH Terms: conditions — Anxiety Disorders; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dance4Healing control group (Active Comparator): Participants will monitor their heart rate for 8 weeks (pre-intervention period), then engage in weekly live zoom dance sessions on digital Dance4Healing platform for 8 consecutive weeks (intervention period), then may elect to continue with monitoring for an additional 12 weeks (3-month post-intervention period for long-term results). During the intervention period, this group will not have a dance buddy.
  Interventions: Behavioral: Dance4Healing Telehealth Live Zoom Sessions
- Dance4Healing Buddy Group (Experimental): Participants will monitor their heart rate for 8 weeks (pre-intervention period), then engage in weekly live zoom dance sessions on digital Dance4Healing platform for 8 consecutive weeks (intervention period), then may elect to continue with monitoring for an additional 12 weeks (3-month post-intervention period for long-term results). During the intervention period, this group will have a dance buddy.
  Interventions: Behavioral: Dance4Healing Telehealth Live Zoom Sessions; Behavioral: Dance Buddy

INTERVENTIONS:
Behavioral: Dance4Healing Telehealth Live Zoom Sessions — Week 1: 2-hour introduction session on Zoom platform with a live dance instructor at the participant's desired level of activity intensity (low, mild, or moderate).
  Weeks 2-8: All participants will be asked to participate in a 1 hour online, instructor-led live class.
Behavioral: Dance Buddy — Following randomization (beginning of intervention period) half of the participants will be assigned a dance "buddy," and will be asked to dance with their buddies using the Dance4Healing TLVP at least 2 additional times/week. This group will have 24/7 access to Dance4Healing Platform during the intervention and post-intervention periods.
  Arms: Dance4Healing Buddy Group

SUMMARY:
This study is to determine if it is feasible to using a Telehealth Dance Platform with patients that have an implantable Cardioverter Defibrillator, and will compare the activity engagement, anxiety, and Quality of Life

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have had an ICD implanted for at least 1 month
2. Patients have access to web-based on-line programs
3. Patient can provide cardiac clearance for exercise from their treating physician OR they have written stress test results from within the last 6 months indicating no ischemia.
4. Patient is 18 years old or greater.

Exclusion Criteria:

1. Patient is non-English speaking.
2. Patient is assessed as having NYHA Class IV heart failure.
3. Patient had ventricular tachycardia (VT), ventricular fibrillation (VF) or has received "tachy" therapy from their ICD within last 4 weeks.
4. Patient has had a change in medical arrhythmia management or ablation procedure within the last 4 weeks.
5. Any medical issues that compromise walking or dancing, including cardiac, neurological or orthopedic .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Activity in hours/day from ICD interrogation as a measure of activity engagement over time | 36 weeks
Change in calculated score from Patient Activation as a measure of Patient Activity Engagement over time | Baseline, Week 8(pre-intervention), Week 16 (post-intervention), Week 28 (long term)
  Scores range from 0-100, higher scores represent higher engagement self reported survey
Total Amount of Time spent accessing the dance platform in minutes as a measure of Activity Engagement during the study intervention | Total time in minutes over the 8 week intervention period
  Total number of minutes that the participant accesses the Dance4Healing platform each week

SECONDARY OUTCOMES:
Change in Anxiety Score over time | Baseline, Week 8(pre-intervention), Week 16 (post-intervention), Week 28 (long term)
  Anxiety will be a calculated score from a 10 question self-reported questionnaire (Florida Shock Anxiety Scale) with a scoring range from 0-50, with higher scores indicating more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Linda K Ottoboni, PhD, Principal Investigator — Stanford Healthcare
Locations (1):
- Stanford Arrhythmia Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No